CLINICAL TRIAL: NCT03538873
Title: "Prevention and Treatment of Depression in the Elderly: A Population-Based Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LLD10446
Record Dates: First submitted 2014-07-07; First posted 2018-05-29 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2018-05

CONDITIONS: Subsyndromic Symptoms of Depression; Subsyndromic Symptoms of Anxiety
Keywords: Subsyndromic symptoms of depression; Subsyndromic symptoms of anxiety; Elderly; Physical activity; Population-based study
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Active Comparator): The assessment of physical activity in the prevention of depression. The intervention program being implemented in this study consists of four steps, lasting three months each:
  Step 1 - Watchful waiting Step 2 - Physical Activity Intervention 1 Step 3 - Physical Activity Intervention 2 Step 4 - Referral to primary care In the case of the CES-D scores remain high, participants will receive orientation to discuss with their doctors the need to receive a specific medication.
  Interventions: Behavioral: Physical activity
- Usual care (No Intervention): Participants in the usual care group will have unrestricted access to usual care for depressive and / or anxiety symptoms.

INTERVENTIONS:
Behavioral: Physical activity
  Arms: Physical activity

SUMMARY:
Considering the rapid increase of the elderly population in Brazil and the growing impact of depression, the third cause of global burden of diseases in the world, the relevance of depression prevention and treatment in older people tend to raise in future years. The investigators planned to screen 2,700 individuals, 60 years and older, from Basic Health Units in the west region of Sao Paulo city, for subsyndromic depressive and / or anxiety symptoms. The elderly will be assessed with a standardized psychiatric interview to calculate the prevalence of subsyndromic symptoms of depression and / or anxiety and the prevalence of depressive and anxiety disorders. Those who do not meet criteria for depressive disorders and / or anxiety will be invited to participate in a randomized clinical trial with 2 arms: a stepped-care prevention program with physical activity (n = 35) or usual care (n = 35). The primary outcome measure will be the cumulative incidence of major depressive disorder, or anxiety disorders, after 12 months.

ELIGIBILITY:
Inclusion Criteria: 60 years or older with subsyndromal symptoms of depression or anxiety, enrolled in one of the selected Project West Region UBS, who agree with the information presented in the free and informed consent term.

A subject is defined as having subsyndromal symptoms of depression and / or anxiety, when he or she scores 13 or more on the CES-D scale, but does not meet criteria for a depressive or anxiety disorder, assessed by applying the "Mini International Neuropsychiatric Interview "(MINI) (Sheehan et al, 1998;. Marques de Azevedo and Zuardi, 2008).

Exclusion Criteria: Those who meet criteria for major depression, dysthymia and / or anxiety disorders, or unable to consent to participate in this research project. All seniors will be interviewed in their homes.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of major depressive disorder, or anxiety disorders | 12 months
  The primary outcome measure will be the cumulative incidence of major depressive disorder, or anxiety disorders after 12 months (MINI, structured interview).

SECONDARY OUTCOMES:
CES-D | 12 months
  Reducing depressive and / or anxiety symptoms, assessed with the CES-D

CONTACTS AND LOCATIONS:
Overall Officials: Cassio MC Bottino, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Institute of Psychiatry, USaoPauloGH, São Paulo, Brazil

REFERENCES:
- [Background] Hunkeler EM, Katon W, Tang L, Williams JW Jr, Kroenke K, Lin EH, Harpole LH, Arean P, Levine S, Grypma LM, Hargreaves WA, Unutzer J. Long term outcomes from the IMPACT randomised trial for depressed elderly patients in primary care. BMJ. 2006 Feb 4;332(7536):259-63. doi: 10.1136/bmj.38683.710255.BE. Epub 2006 Jan 20. PMID 16428253
- [Background] van't Veer-Tazelaar PJ, van Marwijk HW, van Oppen P, van Hout HP, van der Horst HE, Cuijpers P, Smit F, Beekman AT. Stepped-care prevention of anxiety and depression in late life: a randomized controlled trial. Arch Gen Psychiatry. 2009 Mar;66(3):297-304. doi: 10.1001/archgenpsychiatry.2008.555. PMID 19255379
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] de Azevedo Marques JM, Zuardi AW. Validity and applicability of the Mini International Neuropsychiatric Interview administered by family medicine residents in primary health care in Brazil. Gen Hosp Psychiatry. 2008 Jul-Aug;30(4):303-10. doi: 10.1016/j.genhosppsych.2008.02.001. PMID 18585532